CLINICAL TRIAL: NCT02005120
Title: Phase II Study of Intrapleural Administration of Bevacizumab Versus Recombinant Human Endostatin (Endostar) for Refractory Malignant Pleural Effusions in Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Intrapleural Administration of Bevacizumab Versus Endostar for Pleural Effusions in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Chief of Department of Thoracic Oncology, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangUniv
Record Dates: First submitted 2013-11-24; First posted 2013-12-09 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Bevacizumab
  Interventions: Drug: Bevacizumab
- Arm B (Experimental): recombinant human endostatin
  Interventions: Drug: recombinant human endostatin

INTERVENTIONS:
Drug: Bevacizumab — Intrapleural administration of bevacizumab
  Other Names: Avastin
  Arms: Arm A
Drug: recombinant human endostatin — Intrapleural administration of recombinant human endostatin
  Other Names: Endostar
  Arms: Arm B

SUMMARY:
Malignant pleural effusion (MPE) is a common complication of advanced non-small cell lung cancer (NSCLC). Bevacizumab, a humanized monoclonal antibody against vascular endothelial growth factor (VEGF), has been shown to be efficient in suppressing the accumulation of pleural fluid. The other widely used treatment for MPE is recombinant human endostatin.

DETAILED DESCRIPTION:
We designed this clinical trial to determine the efficacy and Safety of intrapleural Bevacizumab versus recombinant human endostatin as a treatment for malignant pleural effusions (MPE) in patients with non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

Patient who was confirmed stage IV NSCLC with malignant pleural effusion confirmed by cytology.

Males or females aged ≥18 years, < 75 years. Eastern Cooperative Oncology Group (ECOG) performance status 0-3. Life expectancy ≥12 weeks. Ability to maintain a drainage catheter. Previous intrapleural administration of chemotherapeutic drugs (preferred bleomycin) Males and females should be contraceptive during the period of the trial until 8 weeks after the last administration of the drug.

Adequate bone marrow, renal, and liver function are required. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Institutional review board-approved informed consent will be obtained for every patient before initiation of any trial-specific procedure or treatment.

Exclusion Criteria:

Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).

Active thoracic cavity or systemic bleeding. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0.

Female subjects should not be pregnant or breast-feeding. Known sensitivity to Bevacizumab or Endostar. Patients must not be on therapeutic anticoagulation with warfarin, heparin or low molecular weight heparin.

Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L.

Adequate renal function: Serum creatinine ≤ 1.5 x ULN, or ≥ 50 ml/min. Adequate liver function :Total bilirubin £ 1.5 x upper limit of normal (ULN) and Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.

Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 12 months

SECONDARY OUTCOMES:
progression free survival (PFS) | 12 months

OTHER OUTCOMES:
Quality of life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Zhao, PhD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (2):
- China (2):
  - Qiong Zhao, Hangzhou, Zhejiang
  - The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang